CLINICAL TRIAL: NCT01660529
Title: A Study of hTERT/Survivin Multi-Peptide Vaccination With Basiliximab And Prevnar For Patients With Metastatic Breast Cancer
Brief Title: Multi-peptide Vaccine With Basilixumab for Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03111
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Subjects with metastatic breast cancer who have failed at least one standard; of care regimen
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hTERT/Survivin Multi-Peptide Vaccination (Experimental): single-arm Phase I study for patients with metastatic breast cancer who have failed at least one regimen for metastatic disease
  Interventions: Biological: hTERT

INTERVENTIONS:
Biological: hTERT

SUMMARY:
Eligible patients will receive subcutaneous vaccinations of the hTERT/survivin/CMV multipeptide vaccine and GM-CSF over a 24 month period. All patients will receive basiliximab 20 mg 1 day prior to the start of vaccinations. Prevnar vaccine will be administered at the time of Vaccines 1,3, and 5. Patients who remain clinically stable after the fourth vaccine, may continue to receive vaccinations every 4 weeks for up to 2 years.

DETAILED DESCRIPTION:
hTERT is widely found in breast cancer cells and has a role in tumor growth and development, making it attractive for immunotherapy. Also, recent data suggest that breast cancer is potentially responsive to immunological therapies. In one trial, patients with advanced cancer received a series of hTERT vaccinations and 4 of 7 patients with advanced breast or prostate carcinoma developed hTERT-specific T lymphocytes. Partial tumor regression was observed in 1 patient. In a second trial, 19 HLA A2+ patients with metastatic breast cancer were vaccinated with hTERT 1540 peptide in adjuvant with GM-CSF. 68% of patients exhibited immunological responses with development of CD8+ hTERT-specific T-cells. Overall survival of vaccine responders was signifiantly better than the overall survival on non-responders. In order to expand the number of possible immune responses and to potentially bypass immune tolerance, multiple peptides have been added to the vaccine. In addition, the monoclonal antibody basiliximab is included to decrease the regulatory T cells which prevent the immune system to work against the tumor, and GM-CSF and Prevnar are used to boost the immune system. Subjects will receive a maximum of 28 vaccinations over a 24 months period.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV (AJCC) breast cancer patients who have failed at least one conventional therapy for metastatic disease.
* HLA-A2 blood positive
* Evidence of measurable or evaluable disease by clinical, radiographic, or laboratory assessment.
* Age greater than 18 years old
* Baseline Eastern Cooperative Oncology Group (ECOG) Clinical Performance Status 0 or 1
* Life expectancy greater than 6 months
* Adequate hematologic function established within 14 days before treatment: WBC equal to or greater than 3.0, Plt equal to or greater than 75,000, Hgb equal to or greater than 10 g/dl
* Adequate renal function established within 14 days before treatment defined as serum creatinine less than 1.5 times upper limit of normal
* Adequate hepatic function established within 14 days before treatment defined as: Total bilirubin, less than 1.5 times upper limit of normal, and ALT and AST less than 2.5 times upper limit of normal
* Contrast CT and/or MRI of the brain negative for central nervous system metastases within 30 days of treatment
* Women of child bearing potential must have a negative pregnancy test (blood or urine) within 14 days before treatment and agree to use appropriate contraception from study screen through the duration of the trial. Men must agree to use appropriate contraception from study screen through the duration of the trial.
* Signed and dated written informed consent

Exclusion Criteria:

* History of brain metastases within the last four years
* Positivity for HIV-1/HIV-2, Hepatitis B virus, and Hepatitis C virus active infection
* The use of the following within 14 days before treatment: Chemotherapy, Radiation therapy, Immunosuppressive drugs, Systemic glucocorticoids, Hematopoietic growth factors, Experimental therapy
* Use of anti-coagulants such as coumadin, heparin, or Lovenox within 14 days before treatment, with the exception of low dose anti-coagulants to maintain intravenous catheter patency.
* Initiation of hormonal agent (such as tamoxifen, anastrazole, or letrozole) in the 30 days before treatment. 6. Patients who have been on a hormonal agent for at least 30 days prior to treatment with progressive or stable disease are permitted to enroll, but required to stay on this hormonal agent for the duration of the study.
* Initiation of immunotherapy (such as trastuzumab-Herceptin) in the 30 days before treatment. Patients who have been on trastuzumab for at least 30 days prior to treatment with progressive or stable disease are permitted to enroll, but required to stay on trastuzumab for the duration of the study.
* History of bone marrow or stem cell transplantation (allogeneic or autologous)
* Pregnant women or nursing mothers
* History of alcohol abuse or illicit drug use within 12 months of study initiation
* Clinically significant comorbid disease or other underlying condition, including major autoimmune disorders that would contraindicate study therapy or confuse interpretation of study results
* Significant psychiatric disorder and any other reason in the Investigators opinion that would jeopardize protocol compliance or compromise the patients ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 1st dose of basiliximab to 30 days after the last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fox, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States